CLINICAL TRIAL: NCT00188513
Title: A Phase I-II Prospective Trial of Conformal Hypofractionated Intensity Modulated Radiotherapy (IMRT) for Localized Adenocarcinoma of the Prostate
Brief Title: Intensity Modulated Radiation Therapy - Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 01-0181-C
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

ARMS (1):
- Conformal intensity modulated radiotherapy (IMRT) (Experimental): All patients shall receive a continuous course of intensity modulated conformal radiotherapy consisting of 66 Gy in 22 (3 Gy) fractions over 4.5 weeks.
  Interventions: Procedure: conformal intensity modulated radiotherapy (IMRT)

INTERVENTIONS:
Procedure: conformal intensity modulated radiotherapy (IMRT)

SUMMARY:
There are several different treatment schedules being used across the world for treatment of prostate cancer with radiation therapy. In order to determine the best radiation treatment for this disease, a study is being performed by the doctors at the Princess Margaret Hospital. This study will try to measure the effectiveness and side effects of an increased dose of radiation to the prostate that is also given over a shorter number of weeks than is usually done. In order to try to reduce the possible side effects of the radiation therapy the treatment will be given using special techniques to shield as much of your normal body tissues as possible. This method of treatment is called conformal intensity modulated radiation therapy, or IMRT.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of adenocarcinoma of the prostate within six months of entry
* Clinical stage T1B, T1C, T2A-C NX MO (see Appendix 1 for staging). Any Gleason score is eligible for entry, but Gleason score must be determined.
* Patients with a PSA >10.0 and Gleason score of 7; or patients with any PSA value and Gleason score of >8 must have clinically negative lymph nodes as determined by a pelvic CT scan done within 12 weeks of entry. A negative bone scan is required before entry for all patients with Gleason score >8, or any patient with a Gleason score of 7, and a PSA >10.
* The patient must not have received any cytotoxic anticancer therapy. Previous or concurrent hormonal therapy for local disease is acceptable.
* ECOG performance status of 1 or less
* Age 80 years old or less
* Serum PSA <25 ng/ml within 4 weeks of study entry
* Informed consent

Exclusion Criteria:

* Patients with history of inflammatory bowel disease or other contraindication to radical radiation therapy
* Patients with prior colorectal surgery
* Any prior pelvic radiotherapy. Any prior TURP done <12 weeks from study entry.
* Any previous cytotoxic chemotherapy
* Patients with prior malignancy except non-melanoma skin carcinoma within 5 years of the diagnosis of prostate cancer

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Estimated)
Dates: Start 2001-05; Primary Completion 2006-04 (Actual); Study Completion 2017-04-04 (Actual)

PRIMARY OUTCOMES:
To determine feasibility and late toxicity of administering 66 Gy in 22 fractions over 4.5 weeks (using conformal IMRT treatment techniques) to the prostate and adjacent tissues in patients with localized prostate ca | at each post treatment follow-up for up to 3 years

SECONDARY OUTCOMES:
To evaluate acute toxicity of therapy | weekly during RT
To evaluate local control as assessed by prostate biopsy at 2.5 years | 2.5 years
To evaluate time to disease progression | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Charles Catton, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada